CLINICAL TRIAL: NCT06782919
Title: Evaluating the Effect of Biofeedback-Based Training on Trunk Neuromuscular Control and Spinopelvic Motion and Loading During Gait in Older Adults With and Without Chronic Low Back Pain
Brief Title: Trunk Control Training and Walking in Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH Funding terminated
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Dennis Anderson, Associate Professor of Orthopedic Surgery, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000980; T32AG023480 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP); Aging
Keywords: Gait; Walking; Neuromuscular control; Wearable Sensors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): For comparison of trunk control and walking between low back pain and health groups.
- Trunk control training (Experimental): Trunk control training is received after baseline measurements in this arm.
  Interventions: Other: Trunk control training

INTERVENTIONS:
Other: Trunk control training — Four sessions of biofeedback trunk movement training, provided once per week.
  Arms: Trunk control training

SUMMARY:
The goal of this observational study and clinical trial is to evaluate control of trunk posture and walking biomechanics in 20 older adults with chronic low back pain and 20 older adult healthy volunteers. A second objective of this study is to evaluate the effect of weekly biofeedback-based trunk control training to control of trunk posture and walking biomechanics. The main question it aims to answer is:

• Does training trunk control improve walking biomechanics in older adults? Researchers will compare older adults with and without chronic low back pain to see if trunk control, walking biomechanics, and the effects of training differ between the groups.

Participants will undergo measurements of trunk control in the laboratory, and of walking in both laboratory and outdoor settings. Trunk training will take place once a week for four weeks, and measurements will be repeated after the training protocol.

ELIGIBILITY:
Inclusion Criteria (Healthy volunteers):

* Men and women, ages 60 - 85 years
* English fluent
* Able to perform activities such as walking, standing, sitting, bending, or lifting without assistance
* Low back pain-free for at least 1 months, characterized by a pain numerical rating scale of <2 (out of 10), and/or <5 (out of 24) on the Roland Morris Disability Questionnaire
* Able to walk without assistance on surfaces of brick, sidewalk, dirt, grass, treadmill, and flat walkway

Inclusion Criteria (Patient group):

* Men and women, ages 60 - 85 years
* English fluent
* Current chronic low back pain (lasting at least 1 months) that care was sought for at BIDMC within the past year.
* Pain numerical rating scale of 2-7 (out of 10) and/or 5-19 (out of 24) on the Roland Morris Disability Questionnaire
* Able to perform activities such as walking, standing, sitting, bending, or lifting without assistance
* Able to walk without assistance on surfaces of brick, sidewalk, dirt, grass, treadmill, and flat walkway

Exclusion Criteria (all subjects):

* Self-reported conditions that might alter spine biomechanics, such as a history of traumatic spine injury or spinal surgery; severe scoliosis which needed brace or surgical treatment; neuromuscular conditions such as Parkinson's disease, hemiplegia, symptomatic spinal stenosis, multiple Sclerosis, or muscular dystrophy.
* Back pain with confirmed diagnosis of underlying diseases or structural anomalies such as rheumatoid arthritis, meningitis, or cancer.
* Severe LBP of greater than 7 (out of maximum 10) on self-report pain VAS. (Subjects otherwise eligible and interested will be followed up weekly and scheduled if LBP subsides to below 7/10 on pain VAS).
* Experienced dizziness, lightheadedness, vertigo, or imbalance within the past three months that occurs frequently (3 times or more) or two or more falls in the past year.
* Use of narcotics
* Latex allergies
* Visual problems that are not corrected by glasses/contact lenses.
* Self-reported recent musculoskeletal injury that is currently severely affecting normal activity or movement. Examples of this could include sprains, strains, dislocations, or fractures that prevent one from walking, standing, sitting, bending, or lifting in a normal manner.
* A score ≥10 on the Short Blessed Test, suggesting possible impaired cognitive function or dementia.
* Two* or more of the following self-reported limits in physical function:

  * Needing help in activities of daily living (ADLs, such as walking across a small room, bathing, toileting, transferring from bed to chair);
  * Unable to walk up and down one flight of stairs without help;
  * Unable to walk half a mile without help.
* Short Physical Performance Battery (SPPB) score <4*

No exclusion criteria shall be based on race, ethnicity, or sex. We will assign subjects to men and women groups for recruitment purposes based on their assigned sex at birth.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Trunk neuromuscular control | Baseline, Training sessions (weekly for 4 weeks), and Followup (approximately week 5, 1 week after training completed).
  Error in performing trunk tracking tasks.
Spinopelvic and lower limb motion | Baseline, and Followup (approximately week 5, 1 week after training completed).
  Joint ranges of motion evaluated during walking
Spinopelvic forces | Baseline, and Followup (approximately week 5, 1 week after training completed).
  Peak and average spine joint compression and shear forces during walking.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E Anderson, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan for sharing in this small preliminary trial; this does not preclude future sharing.